CLINICAL TRIAL: NCT00899665
Title: Proteases in Prostate Cancer Bone Metastasis
Brief Title: Proteases in Patients With Prostate Cancer That Has Spread to the Bone
Status: Completed | Type: Observational
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000483773; P30CA022453 (NIH); WSU-D-2111; WSU-12-35-99(M02)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Anemia; Metastatic Cancer; Myelodysplastic Syndromes; Precancerous Condition; Prostate Cancer
Keywords: stage IV prostate cancer; bone metastases; anemia; monoclonal gammopathy of undetermined significance; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Anemia; Neoplasm Metastasis; Myelodysplastic Syndromes; Precancerous Conditions; Prostatic Neoplasms; Monoclonal Gammopathy of Undetermined Significance | interventions — In Situ Hybridization, Fluorescence; Microarray Analysis; Molecular Diagnostic Techniques; Immunohistochemistry; Biopsy; Radioimmunodetection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: fluorescence in situ hybridization
Genetic: microarray analysis
Genetic: molecular diagnostic method
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: biopsy
Procedure: immunoscintigraphy

SUMMARY:
RATIONALE: Collecting and storing samples of bone marrow and tissue from patients to test in the laboratory may help the study of cancer.

PURPOSE: This laboratory study is comparing proteases (enzymes that break down protein) in patients with prostate cancer that has spread to the bone with patients who do not have cancer that has spread to the bone.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine the roles of proteases and protease-associated molecules in bone metastases in patients with metastatic prostate cancer.

OUTLINE: Patients undergo bone marrow aspiration and core bone biopsies. Tissues are analyzed by immunohistochemistry methods, in situ hybridization assays, gelatin zymography and/or Western blot analysis, and gene profiling analysis in order to visualize and quantitate protease or protease-related levels.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of metastatic prostate cancer

    * Patients with documented bone metastases on radiologic imaging studies must undergo bone marrow biopsy
  * Male patients ≥ 50 years of age without cancer who are scheduled to undergo bone biopsy for other clinically indicated reasons, including any of the following:

    * Myelodysplasia
    * Anemia
    * Monoclonal gammopathy of undetermined significance
  * Male or female patients ≥ 40 years of age without metastatic bone cancer who are scheduled to undergo an orthopedic procedure involving removal of bone specimen

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-07; Primary Completion 2006-09 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Expression and activity of proteases and related molecules

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Cher, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States